CLINICAL TRIAL: NCT03763123
Title: A Phase Ib, Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of Humanized Anti-VEGF Monoclonal Antibody(Sevacizumab) Injection Plus Chemotherapy in Chinese Patients With Platinum-Resistant Recurrent Ovarian Cancer.
Brief Title: A Phase 1b Study of Sevacizumab in Combination With Chemotherapy in Chinese Patients With Platinum-Resistant Recurrent Ovarian Cancer.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM-63-OC-101
Record Dates: First submitted 2018-11-25; First posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sevacizumab +Chemotherapy Combined chemotherapy drug including (Experimental): Investigators selected single-agent chemotherapy on an individual patient basis from the following options, with appropriate premedication according to local standards: paclitaxel 80mg/m2 intravenously (IV)on days 1, 8, 15, and 22 every 4 weeks; or topotecan 4 mg/m2 IV on days 1, 8, and 15 every 4 weeks.
  Interventions: Drug: Sevacizumab; Drug: Paclitaxel; Drug: Topotecan

INTERVENTIONS:
Drug: Sevacizumab — Drug: Sevacizumab escalating doses of Sevacizumab : 0.5mg/kg，1mg/kg，1.5mg/kg and 2mg/kg
Drug: Paclitaxel — paclitaxel 80mg/m2 as a > 3-hour IV infusion on days 1, 8,15, and 22 every 4 weeks;
Drug: Topotecan — topotecan 4 mg/m2 as a >30 minute IV infusion on days 1, 8, and 15 every 4 weeks ;

SUMMARY:
This is an open-label, multicenter, dose-escalation study designed to assess the safety, tolerability, and pharmacokinetics of Humanized Anti-VEGF Monoclonal Antibody (Sevacizumab) Injection in combination with Chemotherapy in Chinese patients with Platinum-Resistant Recurrent Ovarian Cancer. This study includes two stages. Stage 1 is the dose-escalation stage. Once the maximum tolerated dose (MTD of Sevacizumab has been established, additional patients will be enrolled in the cohort-expansion stage (Stage 2).

DETAILED DESCRIPTION:
This is an open-label, multicenter, dose-escalation study designed to assess the safety, tolerability, and pharmacokinetics of Humanized Anti-VEGF Monoclonal Antibody (Sevacizumab) Injection in combination with Chemotherapy in Chinese patients with Platinum-Resistant Recurrent Ovarian Cancer. This study includes two stages. Stage 1 is the dose-escalation stage. Once the maximum tolerated dose (MTD of Sevacizumab has been established, additional patients will be enrolled in the cohort-expansion stage (Stage 2).

ELIGIBILITY:
Inclusion Criteria:

1. age≥18 years
2. Histologically documented platinum resistant
3. EOC, FTC, or PPC of the following types: adenocarcinoma not otherwise specified (NOS), clear cell adenocarcinoma, endometriod adenocarcinoma, malignant Brenner's tumor, mixed epithelial carcinoma, mucinous adenocarcinoma, serous adenocarcinoma, transitional cell carcinoma and undifferentiated carcinoma.
4. At least one measurable leision. (according to RECIST 1.1 )
5. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1.
6. Adequate hematologic function: ANC ≥ 1.5 × 10^9 /L, HB ≥ 90 g /L (blood transfusion allowed), PLT ≥ 100 ×10^9 /L; Adequate hepatic function: ALT ≤ 2.5 × ULN, AST ≤ 2.5 × ULN, TBIL ≤ 1.5 × ULN (patients with liver metastases ALT ≤ 5 × ULN, AST ≤ 5 × ULN); Adequate renal function: creatinine ≤ 1 × ULN; Coagulation function: INR ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN
7. Progression within 6 months from completion of a minimum of 4 platinum therapy cycles.
8. Life expectancy ≥12 weeks.
9. At least 4 weeks from the last chemotherapy. If patients received anti-tumor biological products, at least four t1/2 of washout period is needed
10. Toxicity from previous treatment has to restore to ≤ grade 1 (NCI CTC4.0)
11. Patients signed written inform consent.
12. Willingness and capability to communicate with investigators and to comply with protocol requirements

Exclusion Criteria:

1. Previous treatment with > 2 anti-cancer regimens.
2. Patients whose disease was refractory to their previous platinum treatment. (Refractory disease was defined as those patients who progressed during the preceding platinum treatment.)
3. Ovarian tumors with low malignant potential (i.e. borderline tumors).
4. Patients with a prior invasive malignancy (except non-melanoma skin cancer) or whose prior malignancy treatment contraindicated the current protocol therapy.
5. Any prior radiotherapy to the pelvis or abdomen.
6. Patients with serious non-healing wound, ulcer, or bone fracture.
7. patients with a history of bowel obstruction (including subocclusive disease) related to underlying disease, a history of abdominal fistula, GI perforation, or intra-abdominal abscess or evidence of rectosigmoid involvement by pelvic examination, bowel involvement on computed tomography, or clinical symptoms of bowel obstruction.
8. Serious infection requiring intravenous antibiotic therapy
9. history or evidence of thrombotic or hemorrhagic disorder within 6 months before first study treatment
10. untreated CNS disease unrelated to cancer or symptomatic CNS metastasis
11. Patients with clinically significant cardiovascular disease. This included:Uncontrolled hypertension, defined as systolic > 150 mmHg or diastolic > 90 mmHg;Myocardial infarction or unstable angina > 6 months prior to registration;New York Heart Association (NYHA) Grade II or greater congestive heart failure;Serious cardiac arrhythmia requiring medication. This did not include asymptomatic, atrial fibrillation with controlled ventricular rate.
12. left ventricular ejection fraction below the institutional lower limit of normal
13. pre-existing neuropathy ≥ CTC Grade 2 for those in the paclitaxel group
14. Known allergies to any excipient in the study drug
15. Pregnant and lactating women
16. Patients with proteinuria (urine protein >1+ at screening, or urine protein 1+, not recover to normal value within 24h)
17. Previously received anti-VEGF protein drugs, such as Bevacizumab, Sevacizumab
18. Patients with or with anticipation of invasive procedures as defined below:Major surgical procedure or significant traumatic injury within 28 days prior to the first date of sevacizumab therapy;Major surgical procedure anticipated during the course of the study. This included, but was not limited to abdominal surgery (laparotomy or laparoscopy) prior to disease progression;Core biopsy, within 7 days prior to randomization.
19. Participation in other clinical trials within 4 weeks before enrollment
20. The investigators consider the patients are not suitable for this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 3 years
The ratio of adverse of event | 3 years

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | 3 years
  Maximum Plasma Concentration [Cmax]
Area Under the Curve [AUC], | 3 years
  Area Under the Curve [AUC]
Tmax | 3 years
  Tmax for Cmax of sevacizumab
Objective Response Rate (ORR) | 3 years
Disease Control Rate (DCR) | 3 years
Overall Survival (OS) | 3 years
Progression Free Survival (PFS) | 3 years

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The first affiliated hospital,sun yat-sen university, Guangzhou, Guangdong
  - the Affiliated Cancer Hospital of Harbin Medical University, Harbin, Hei Longjiang
  - Hunan Cancer Hospital, Changsha, Hunan
  - Wuhan Union Hospital, Wuhan, Hunan

IPD SHARING:
Plan to Share IPD: No